CLINICAL TRIAL: NCT04320875
Title: Stimulate Brain to Reduce Pain Among Patients With Knee Osteoarthritis
Brief Title: Stimulate Brain and Reduce Knee Pain Due to Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMDU/IEC/108P; U1111-1249-2403 (Other: Universal Trial Number (UTN) by WHO ICTRP)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis
Keywords: Transcranial direct current stimulation; Pain; knee osteoarthritis; Exercise therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Transcranial Direct Current Stimulation; 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial direct current stimulation (tDCS) group (Experimental): Fourty patients with KOA will receive structured tDCS (MA-tDCS, Walnut-Medical, Johnstown, PA) treatment. Two pair of sponge electrodes soaked with saline and fixed to head with elastic bands. The transcranial direct current stimulation will be applied by a constant current device with an intensity of 2mA
  Interventions: Other: Transcranial direct current stimulation
- Conventional Physiotherapy (CPT) group (Active Comparator): Individual with KOA will be educated on how to do the set of exercises correctly at their home during the first session. Consisted of nine exercises including muscle strengthening and flexibility training.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Transcranial direct current stimulation — Anode electrode -C3/C4 (International 10-20 electroencephalogram system), contralateral side of the most affected knee) Cathode electrode- contralateral supraorbital area. 2 mA intensity for 20 minutes, one session/day for 3 days/week for 8 weeks)
  Other Names: tDCS
  Arms: Transcranial direct current stimulation (tDCS) group
Other: Conventional Physiotherapy — 1. Warm-up exercises: Walking at the usual speed on a flat surface for 10 min ( 3sets X10 Reps X 3 min rest in between)
  2. Hamstring and calf gentle stretches. ( 3sets X10 Reps X 3 min rest in between)
  3. Straight leg raise (SLR) ( 3sets X10 Reps X 3 min rest in between)
  4. Quadriceps setting ( 3sets X10 Reps X 3 min rest in between)
  5. Pillow squeeze ( 3sets X10 Reps X 3 min rest in between)
  6. Heel raise ( 3sets X10 Reps X 3 min rest in between)
  7. One leg balance ( 3sets X10 Reps X 3 min rest in between)
  8. Step ups ( 3sets X10 Reps X 3 min rest in between)
  9. Quadriceps strengthening exercises ( 3sets X10 Reps X 3 min rest in between)
  Other Names: CPT
  Arms: Conventional Physiotherapy (CPT) group

SUMMARY:
Osteoarthritis (OA) knee is chronic, slowly progressive, degenerative disease of joint which affects articular cartilage and accompanied by pain, swelling and loss of function . OA is often considered as the serious joint disease as it has negative impact on quality of life among elderly population, it is the major cause for the reduced mobility. At cental level, due to imbalance in endogenous pain modulation there is reduce capacity of brain to inhibit the pain. Therefore, dysregulation in the central modulation of pain further leads to maladaptive changes in the brain structure. Transcranial direct current stimulation is a non-invasive method to modulate the brain structure by using a week direct current applied through the scalp in painless way. Multi-session for prolonged time can induce neuroplastic changes in the brain.

The aim of the study is to demonstrate the effectiveness of tDCS in reducing the pain among patients with chronic knee OA and to modulate the plastic changes in brain structure.

A total of 80 patients with KOA will be recruited by the convenience sampling to participate in this two group pretest-posttest, double blinded randomized clinical study. After the demographics, recruited 80 patients with KOA will be randomly divided into two groups, transcranial direct current stimulation (tDCS) group and conventional physiotherapy (CPT) group with by block randomization. Patients with KOA in tDCS group will be provided with Active tDCS and conventional physiotherapy and CPT group will receive structured exercises protocol. Pre-post changes in the outcome measures will be documented at baseline and end of 8-week post intervention. Each session will last for approximately 30 minutes duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with clinical knee OA according to the diagnostic criteria of ACR were included in the study

Exclusion Criteria:

* Unwillingness to participate in the study
* Recent history (within the last 3 months) of physical therapy to the same joint
* Recent history (within the last 3 months) of intra-articular procedure (injection and/or lavage) to the knee
* History of knee surgery/fracture
* Acute synovitis/arthritis including the infectious conditions
* Taking pain relief medications
* Any metal implantation near site of stimulation

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Digitalized pain pressure algometer (ALGO-DS-01) | Changes will be measured at baseline and end of 8 week intervention
  Pain intensity will be measured using calibrated digitalized pain pressure algometer (ALGO-DS-01) in patients with KOA.

SECONDARY OUTCOMES:
Western Ontario and Mc Master Universities Osteoarthritis Index (WOMAC) | Changes will be measured at baseline and end of 8 week intervention
  The Western Ontario and Mc Master Universities Osteoarthritis Index (WOMAC) will be used to evaluate the disease-specific self-reported symptoms of OA. This form is comprised of 24 questions in three categories including pain (5 questions), stiffness (2 questions), and physical function (17 questions)

CONTACTS AND LOCATIONS:
Overall Officials: Asir J Samuel, Ph.D, Principal Investigator — Maharishi Markandeshwar Medical College and Hospital; Adarsh K Srivastav, MPT, Study Director — Maharishi Markandeshwar Medical College and Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahn H, Woods AJ, Kunik ME, Bhattacharjee A, Chen Z, Choi E, Fillingim RB. Efficacy of transcranial direct current stimulation over primary motor cortex (anode) and contralateral supraorbital area (cathode) on clinical pain severity and mobility performance in persons with knee osteoarthritis: An experimenter- and participant-blinded, randomized, sham-controlled pilot clinical study. Brain Stimul. 2017 Sep-Oct;10(5):902-909. doi: 10.1016/j.brs.2017.05.007. Epub 2017 May 19. PMID 28566193
- [Result] Srivastav AK, Sharma N, Samuel AJ. tDCS combined with cognitive training in a patient with chronic traumatic head injury. Neurophysiol Clin. 2020 Apr;50(2):133-134. doi: 10.1016/j.neucli.2020.02.004. Epub 2020 Mar 5. No abstract available. PMID 32147282
- [Result] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Result] Lluch E, Torres R, Nijs J, Van Oosterwijck J. Evidence for central sensitization in patients with osteoarthritis pain: a systematic literature review. Eur J Pain. 2014 Nov;18(10):1367-75. doi: 10.1002/j.1532-2149.2014.499.x. Epub 2014 Apr 3. PMID 24700605